CLINICAL TRIAL: NCT01947218
Title: EFFECT OF SMOKING ON MUCUS HYPERSECRETION MECHANISMS IN ASTHMA AND CHRONIC OBSTRUCTIVE PULMONARY DISEASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013-A00553-42; 2013-14 (Other: AP HM)
Record Dates: First submitted 2013-08-01; First posted 2013-09-20 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: CHRONIC OBSTRUCTIVE PULMONARY DISEASE (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (4):
- smoking COPD (Experimental)
  Interventions: Procedure: bronchial biopsies; Other: Determination of CO in exhaled air
- smoking without COPD (Experimental)
  Interventions: Procedure: bronchial biopsies; Other: Determination of CO in exhaled air
- No Smoking Control (Other)
  Interventions: Procedure: bronchial biopsies; Other: Determination of CO in exhaled air
- severe asthma (Experimental)
  Interventions: Procedure: bronchial biopsies; Other: Determination of CO in exhaled air

INTERVENTIONS:
Procedure: bronchial biopsies
Other: Determination of CO in exhaled air

SUMMARY:
Asthma and COPD are characterized by an accelerated decline in lung function associated with incompletely reversible airflow obstruction. This could be the result of lung structural changes and inflammation. Tissue repairing mechanisms may result in a restitution ad integrum of bronchial epithelium. But in most cases, especially in COPD and severe asthma, the "remodeling" is characterized by mucus cells hyperplasia, overproduction of mucus, and physicochemical, biological and immunological changes. Clinically, this mucus overproduction is reported by patients as the clinical symptom called "chronic bronchitis". Generally, it develops at a bronchiolar level where it is responsible for the progression of these diseases. There is a paradox, because the intrinsic properties of mucus seem rather beneficial so fighting against it may not be really wise at long-term. Especially its defensive effect against microbial agents which remains poorly explained. Currently, no treatment aims to reduce the production of mucus and mechanisms leading to such an overproduction are poorly understood in severe asthma and COPD. The identification of new targets to treat this overproduction of mucus in COPD is therefore of major interest.

In view of current knowledge, inflammatory mediators and signal transduction leading to increased mucin production and increased number of goblet cells are probably IL-9, IL-13, IL -1ß and TNF-α involving calcium-sensitive chloride channels. Intracellular signaling pathways seem to be based on STAT-6, FOXA2, SPDEF, EGFR and / or COX-2

ELIGIBILITY:
Inclusion Criteria:

* The patient must be given free and informed consent and signed the consent
* The patient must be a member or beneficiary of a health insurance plan
* Women and men are included (s)
* The patient is aged at least 18 years

Exclusion Criteria:

* neoplastic disease extent
* Other progressive lung disease (tuberculosis, diseases of the pulmonary interstitium, active or recent pulmonary infection.)
* Patient unstable or had experienced exacerbation in the previous month study.
* Unable to understand the nature and purpose of the study
* Not affiliated to the French social security
* Making their military or military service career
* During periods of exclusion on another protocol
* Patients who are mentally or legally can not give consent.
* Patients with recent psychiatric disorders (less than a year).
* The illicit drugs or alcohol.
* Pregnant women, nursing mothers and women in labor;
* Women of childbearing potential without effective contraception (specified in the protocol)
* Persons deprived of their liberty by a judicial or administrative decision, hospitalized without consent and persons admitted to a health or social establishment for purposes other than research;
* Minors;
* The adults subject to a measure of legal protection or unable to consent;
* The people in emergency situations can not give consent.
* People with a cons-indication for bronchial biopsies (coagulation disorders, anticoagulation can be suspended ...)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
measure the impact of cigarette smoke on the formation and composition of mucus produced by the bronchial epithelium | 4 years
  (physicochemical properties, protein composition and potentially beneficial role in innate immunity)

SECONDARY OUTCOMES:
measure the concentration of intracellular calcium | 4 years
  induced by cigarette smoke measured by confocal microscopy using a fluorochrome (Fura-2)

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France